CLINICAL TRIAL: NCT04785391
Title: A Sample Collection Study to Validate the NEPHROCLEAR™ CCL14 Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Astute Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Diamond
Record Dates: First submitted 2021-03-01; First posted 2021-03-05 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Patients with KDIGO stage 2 or 3 AKI
  Interventions: Diagnostic Test: Urine collection for NEPHROCLEAR CCL14 Test

INTERVENTIONS:
Diagnostic Test: Urine collection for NEPHROCLEAR CCL14 Test — Urine will be collected and banked for future analysis with the NEPHROCLEAR CCL14 Test

SUMMARY:
The objective of this sample collection study is to collect urine samples to validate the NEPHROCLEAR™ CCL14 Test in patients with KDIGO stage 2 or 3 AKI. This study is observational and will have no impact on the medical management of the subject.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 21 years of age or older;
2. Receiving care in an intensive care unit;
3. Expected to remain in the ICU for at least 48 hours after enrollment;
4. Use of indwelling urinary catheter as standard care at the time of enrollment;
5. Subject must have acute kidney injury (KDIGO Stage 2 or Stage 3) at the time of sample collection;
6. Urine sample must be collected within 36 hours of meeting KDIGO Stage 2 criteria;
7. Written informed consent provided by patient or legally authorized representative (LAR).

Exclusion Criteria:

1. Prior kidney transplantation;
2. Comfort-measures-only status;
3. Already receiving dialysis (either acute or chronic) or in imminent need of dialysis at the time of enrollment;
4. Known infection with human immunodeficiency virus (HIV) or active hepatitis (acute or chronic);
5. Special populations, pregnant women, prisoners or institutionalized individuals.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients with KDIGO stage 2 or 3 AKI.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Persistent Severe Acute Kidney Injury as Determined by Physician Adjudication | Within 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Jay L Koyner, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States